CLINICAL TRIAL: NCT06559202
Title: Evaluation of Inguinal and Axillary Lymph Node Size Distribution for Safe Intralymphatic Injection
Brief Title: Inguinal and Axillary LN Size Distribution
Status: Completed | Type: Observational
Sponsor: Gachon University Gil Medical Center (Other)
Collaborators: Dankook University (Other)
Responsible Party: Principal Investigator, Sangmin Lee, MD, Professor, Gachon University Gil Medical Center
Other Study IDs: GDIRB2024-098
Record Dates: First submitted 2024-08-10; First posted 2024-08-19 (Actual); Last update posted 2024-08-19 (Actual); Status verified 2024-08

CONDITIONS: Lymph Nodes
Keywords: lymph nodes; immunotherapy; intralymphatic immunotherapy; computed tomography

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- CT group: Participants who underwent chest and abdominopelvic computed tomography on the same day for health screening purposes
  Interventions: Diagnostic Test: chest and abdominoplevic CT

INTERVENTIONS:
Diagnostic Test: chest and abdominoplevic CT — chest and abdominopelvic computed tomography on the same day for health screening purposes

SUMMARY:
Recently, intralymphatic allergen-specific immunotherapy (ILIT) showed promising treatment outcomes for allergic rhinoconjunctivitis. However, the normal size distribution of superficial lymph nodes (LNs) on the trunk that are potential target LNs for ILIT has not been evaluated.

The objective of this study is to investigate the distribution of LN size in inguinal and axillary area.

DETAILED DESCRIPTION:
In this study, the long-axis diameters of the largest LNs in the inguinal and axillary areas were retrospectively measured in subjects who underwent chest and abdominopelvic computed tomography on the same day for health screening purposes from September 2022 to November 2022.

ELIGIBILITY:
Inclusion Criteria:

* subjects who underwent chest and abdominopelvic computed tomography on the same day for health screening purposes

Exclusion Criteria:

* Malignancy
* Follow-up less than 1-year

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: subjects who underwent chest and abdominopelvic computed tomography on the same day for health screening purposes
Sampling Method: Non-Probability Sample
Enrollment: 133 (Actual)
Dates: Start 2022-09-02 (Actual); Primary Completion 2022-11-30 (Actual); Study Completion 2022-11-30 (Actual)

PRIMARY OUTCOMES:
Inguinal LN size | On the day when chest and abdominopelvic CT was performed during the study period from 1st SEP 2022 to 30th NOV 2022
  The long-axis diameter of the largest inguinal lymph node
Axillary LN size | On the day when chest and abdominopelvic CT was performed during the study period from 1st SEP 2022 to 30th NOV 2022
  The long-axis diameter of the largest axillary lymph node

SECONDARY OUTCOMES:
Subjects with inguinal LN size ≥ 10mm | On the day when chest and abdominopelvic CT was performed during the study period from 1st SEP 2022 to 30th NOV 2022
  The number of subjects in whom the long-axis diameter of the largest inguinal lymph node is 10 mm or more.
Subjects with axillary LN size ≥ 10mm | On the day when chest and abdominopelvic CT was performed during the study period from 1st SEP 2022 to 30th NOV 2022
  The number of subjects in whom the long-axis diameter of the largest axillary lymph node is 10 mm or more.

OTHER OUTCOMES:
Correlation between inguinal and axillary LN sizes | On the day when chest and abdominopelvic CT was performed during the study period from 1st SEP 2022 to 30th NOV 2022
  Correlation between the long-axis diameter of the largest LNs in inguinal area and those in axillary area
Correlation between inguinal LN size and age | On the day when chest and abdominopelvic CT was performed during the study period from 1st SEP 2022 to 30th NOV 2022
  Correlation between the long-axis diameter of the largest inguinal LN and age
Correlation between axillary LN size and age | On the day when chest and abdominopelvic CT was performed during the study period from 1st SEP 2022 to 30th NOV 2022
  Correlation between the long-axis diameter of the largest axillary LN and age
Correlation between inguinal LN size and height | On the day when chest and abdominopelvic CT was performed during the study period from 1st SEP 2022 to 30th NOV 2022
  Correlation between the long-axis diameter of the largest inguinal LN and height
Correlation between axillary LN size and height | On the day when chest and abdominopelvic CT was performed during the study period from 1st SEP 2022 to 30th NOV 2022
  Correlation between the long-axis diameter of the largest axillary LN and height
Correlation between inguinal LN size and BMI | On the day when chest and abdominopelvic CT was performed during the study period from 1st SEP 2022 to 30th NOV 2022
  Correlation between the long-axis diameter of the largest inguinal LN and BMI
Correlation between axillary LN size and BMI | On the day when chest and abdominopelvic CT was performed during the study period from 1st SEP 2022 to 30th NOV 2022
  Correlation between the long-axis diameter of the largest axillary LN and BMI
Correlation between inguinal LN size and weight | On the day when chest and abdominopelvic CT was performed during the study period from 1st SEP 2022 to 30th NOV 2022
  Correlation between the long-axis diameter of the largest inguinal LN and weight
Correlation between axillary LN size and weight | On the day when chest and abdominopelvic CT was during the study period from 1st SEP 2022 to 30th NOV 2022
  Correlation between the long-axis diameter of the largest axillary LN and weight

CONTACTS AND LOCATIONS:
Overall Officials: So Hyun Park, MD, PhD, Study Director — Gachon University Gil Medical Center
Locations (1):
- Gachon University Gil Medical Center, Incheon, South Korea

IPD SHARING:
Plan to Share IPD: No
I think that IPD of this observational retrospective mono-center pilot study needs not be shared.